CLINICAL TRIAL: NCT02775006
Title: A Randomized Phase III Study of Docetaxel Versus Intercalated Erlotinib Docetaxel Combination Therapy in Patients With Relapsed EGFR (Epidermal Growth Factor Receptor) Wild Type, ALK(Anaplastic Lymphoma Kinase) Negative Non Squamous Cell Carcinoma. (NVALT 18 Study)
Brief Title: Docetaxel Versus Intercalated Erlotinib-docetaxel in Patients With Relapsed EGFR Wild Type, ALK Negative Non Squamous Cell Carcinoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: accrual to slow, target not achievable
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Dutch Society of Physicians for Pulmonology and Tuberculosis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NVALT 18
Record Dates: First submitted 2016-04-12; First posted 2016-05-17 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Carcinoma, Non-small Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docetaxel (Active Comparator): Docetaxel 75mg/m2 every 21 days until disease progression or toxicity related
  Interventions: Drug: Docetaxel
- Docetaxel plus erlotinib (Active Comparator): Docetaxel 75mg/m2 on Day 1 plus erlotinib 150mg/day days 2-16, every 21 days, until disease progression, or toxicity related.
  Interventions: Drug: Docetaxel; Drug: Erlotinib

INTERVENTIONS:
Drug: Docetaxel — 75mg/m2
  Other Names: Taxotere
Drug: Erlotinib — 150mg/day
  Other Names: Tarceva
  Arms: Docetaxel plus erlotinib

SUMMARY:
The objective of this study is to investigate the effect of docetaxel monotherapy and the combination of docetaxel intercalated erlotinib in patients with relapsed EGFR wild type, ALK negative non squamous cell carcinoma.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effect of docetaxel monotherapy and the combination of docetaxel intercalated erlotinib in patients with relapsed EGFR wild type, ALK negative non squamous cell carcinoma.

As pemetrexed is standard first line treatment, the combination of erlotinib docetaxel in non-squamous NSCLC should be investigated as second line treatment. Also the question has to be answered whether the combination outperforms monotherapy treatments.

After stratification for ECOG-performance status (0-1), response to prior treatment (CR, PR, SD versus PD), treatment free interval after platinum based therapy (<6 months versus >6 months) and maintenance, patients will be centrally randomized to receive either docetaxel (arm A) or docetaxel plus erlotinib (arm B).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed EGFR wild type, ALK negative, non-squamous cell carcinoma, locally advanced and metastatic disease stage IIIB and IV. Evidence of disease progression after one cytotoxic treatment platinum containing regimen. Immunotherapy pretreatment is allowed
2. Complete recovery from prior chemotherapy side effects to < Grade 2.
3. At least one unidimensionally measurable lesion meeting RECIST criteria.
4. ECOG PS 0-1.
5. Age ≥ 18 years.
6. Adequate organ function, including:

   * Adequate bone marrow reserve: ANC > 1.5 x 109/L, platelets ≥ 100 x 109/L.
   * Hepatic: bilirubin ≤1.5 x ULN (upper limit normal), AP, ALT, AST ≤ 1.5 x ULN. AP, ALT, and AST ≤5 x ULN is acceptable if the liver has tumor involvement.
   * Renal: calculated creatinine clearance ≥ 40 ml/min based on the Cockcroft-Gault formula.
7. Male and female patients with reproductive potential must use an approved contraceptive method, if appropriate. Female patients with childbearing potential must have a negative serum pregnancy test within 7 days prior to study enrollment.
8. Signed informed consent.
9. Patient compliance and geographical proximity that allow adequate follow up.
10. Patients who have undergone cranial irradiation for brain metastases more than 4 weeks before inclusion in our protocol, provided that they are clinically fit to undergo second line treatment

Exclusion Criteria:

1. Pregnant or lactating women.
2. Patients with medical risks because of non-malignant disease as well as those with active uncontrolled infection.
3. Documented brain metastases unless the patient has completed local therapy for central nervous system metastases at least 4 weeks before enrollment and has been off corticosteroids for at least two weeks before enrollment. Prophylactic irradiation at least 4 weeks prior to enrollment is accepted.
4. Maintenance treatment with erlotinib or other TKI (Tyrosine Kinase Inhibitor), or docetaxel. Maintenance treatment with pemetrexed is allowed. Previous treatment with an EGFR-TKI or docetaxel within 6 months prior to enrollment.
5. Inability or unwillingness to take dexamethasone.
6. Concomitant treatment with any other experimental drug under investigation.
7. Patients experiencing disease progression within 2 months after the start of platinum based chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-10-14 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
progression free survival | from the date of randomization to the first date of progression of disease or of death from any cause up to 24 months after last treatment administration

SECONDARY OUTCOMES:
quantitative and qualitative adverse events | from the date of randomization until resolution or stabilization of the event and up to 30 days after the last study medication/treatment
  Adverse events will be graded according to NCI Common Toxicity Criteria version 4.03
response rates | Every six weeks from date of randomization until the date of first documented progression or date of death from any cause up to 24 months after last treatment administration
duration of response | from the date of the first objective status assessment of a complete or partial response to the first date of progression of disease or death from any cause up to 24 months after last treatment administration
overall survival | from the date of randomization to the date of death from any cause up to 24 months after last treatment administration
  Evaluation of overall survival (OS)

OTHER OUTCOMES:
Erlotinib dose level variance in blood | Every six weeks from randomisation up until last treatment administration (up until 48 weeks)
  Therefore in patients on erlotinib every 6 weeks through dose levels in blood will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Joachim G Aerts, MD PhD, Principal Investigator — Dutch Society of Physicians for Pulmonology and Tuberculosis
Locations (19):
- Netherlands (19):
  - VUmc Medical Center, Amsterdam, North Holland
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - Gelre Ziekenhuis, Apeldoorn
  - Amphia Hospital, Breda
  - Albert Schweitzer ziekenhuis, Dordrecht
  - Ziekenhuis Gelderse Vallei, Ede
  - Maxima Medisch Centrum, Eindhoven
  - Martini Ziekenhuis, Groningen
  - Spaarne Gasthuis, Hoofddorp
  - MCL, Leeuwarden
  - Maastricht University Medical Center, Maastricht
  - Laurentius Hospital, Roermond
  - St. Fransicus Gasthuis, Rotterdam
  - Ikazia, Rotterdam
  - Erasmus MC, Rotterdam
  - Haga, The Hague
  - Medical Center Haaglanden, The Hague
  - St. Antonius ziekenhuis, Utrecht
  - VieCuri Medisch Centrum voor Noord-Limburg, Venlo

IPD SHARING:
Plan to Share IPD: No